CLINICAL TRIAL: NCT00370552
Title: A Phase II Open Label, Randomized, 3 Arm Trial of 2 Schedules of Ixabepilone Plus Bevacizumab and Paclitaxel Plus Bevacizumab as First Line Therapy for Locally Recurrent or Metastatic Breast Cancer
Brief Title: A Trial of 2 Schedules of Ixabepilone Plus Bevacizumab and Paclitaxel Plus Bevacizumab for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-115
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Bevacizumab; Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg (Experimental)
  Interventions: Drug: Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg
- Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg (Experimental)
  Interventions: Drug: Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg
- Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg (Active Comparator)
  Interventions: Drug: Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg

INTERVENTIONS:
Drug: Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg — Ixabepilone,16 mg/m^2, administered as a 1-hour intravenous (IV) infusion on Days 1, 8, and 15 of a 28-day cycle until disease progression or unacceptable toxicity. Bevacizumab, 10 mg/kg, administered as IV infusion every 2 weeks. Bevacizumab to be infused over 90 minutes for the first dose, and if well tolerated for 60 minutes, for the second dose. Then if still tolerated, over 30 minutes for subsequent infusions. Bevacizumab was to be dosed until disease progression or unacceptable toxicity.
  Other Names: IXEMPRA; BMS-247550
  Arms: Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg
Drug: Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg — Ixabepilone, 40 mg/m^2, administered as a 3-hour IV infusion on Day 1 of a 21-day cycle until disease progression or unacceptable toxicity (After Cycle 4, dose reduction to 32 mg/m^2 was to be implemented for all subsequent cycles.) Bevacizumab, 15 mg/kg, administered as IV infusion every 3 weeks. Bevacizumab to be infused over 90 minutes for the first dose, and if well tolerated for 60 minutes, for the second dose. Then if still tolerated, over 30 minutes for subsequent infusions. Bevacizumab was to be dosed until disease progression or unacceptable toxicity.
  Other Names: IXEMPRA; BMS-247550
  Arms: Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg
Drug: Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg — Paclitaxel, 90 mg/m^2, given as a 1-hour IV infusion on Days 1, 8, and 15 of a 28-day cycle until disease progression or unacceptable toxicity. Bevacizumab, 10 mg/kg, administered as IV infusion every 2 weeks. Bevacizumab infused over 90 minutes for the first dose, and if well tolerated, over 60 minutes for the second dose. If still tolerated, over 30 minutes for subsequent infusions. Bevacizumab was to be dosed until disease progression or unacceptable toxicity.
  Other Names: TAXOL; BMS-181339
  Arms: Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg

SUMMARY:
The purpose of this clinical research study is to learn if ixabepilone plus bevacizumab is effective in shrinking or stopping the growth of cancer when given as first-line chemotherapy in participants with metastatic breast cancer. The study will also assess the safety of this combination treatment.

ELIGIBILITY:
Inclusion criteria:

* Locally recurrent or metastatic breast cancer, previously untreated with chemotherapy for advanced disease.
* At least 1 target lesion per RECIST criteria. Locally recurrent disease must not be amenable to resection with curative intent.
* No previous cytotoxic chemotherapy for locally recurrent/metastatic disease.
* Relapse 12 months or more after completing prior adjuvant or neoadjuvant taxane therapy.
* No previous breast cancer known to overexpress or amplify the human epidermal growth factor receptor 2 gene.
* Prior hormonal therapy in adjuvant, recurrent, or metastatic setting allowed but must have been discontinued at least 2 weeks before randomization.
* Karnofsky performance status of 80 to 100 or Eastern Cooperative Oncology Group performance status of 0 to 1.
* Estimated life expectancy of at least 12 weeks.
* Recovery from recent therapy (except for alopecia), including chemotherapy, immunotherapy, biologic therapy, or investigational product. Any such therapy must have been completed at least 3 weeks before randomization and at least 6 weeks from use of nitrosourea, or mitomycin.
* Recovery from recent surgery and radiation therapy. At least 1 week since minor surgery and/or focal/palliative radiation therapy; at least 3 weeks from radiation; at least 4 weeks from major surgery; and at least 8 weeks from liver resection, thoracotomy, or neurosurgery.
* Absolute neutrophil count ≥1500/mm^3.
* Hemoglobin ≥9 g/dL.
* Platelets ≥100,000/mm^3.
* Total bilirubin ≤1.5 times the upper limit of normal (ULN).
* Aspartate aminotransferase or alanine aminotransferase ≤2.5*ULN.
* Normal partial thromboplastin time and either international normalized ratio or prothrombin time <1.5*ULN.
* Serum creatinine ≤1.5*ULN or 24-hour creatinine clearance >60 mL/min.
* Urine dipstick for proteinuria <2+ (negative, trace, or +1). Participants with ≥2+ proteinuria at baseline were to undergo 24-hour urine collection and demonstrate ≤1g of protein in 24 hours to be eligible.

Exclusion criteria:

* Women of child-bearing potential (WOCBP) unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and up to 6 months after treatment with bevacizumab.
* Women who were pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Sexually active fertile men, whose partners were WOCBP, not using an adequate method of birth control.
* Evidence of baseline sensory or motor neuropathy.
* Serious infection or nonmalignant medical illnesses uncontrolled or the control of which could be jeopardized by this therapy.
* History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, serious gastric ulcer, or bone fracture within 6 months of study entry.
* History of hypertensive crisis or hypertensive encephalopathy.
* Significant vascular disease.
* Clinically significant cardiovascular disease.
* Baseline left ventricular ejection fraction by multiple-gated acquisition scan or echocardiogram for subjects with prior exposure to anthracyclines not within institutional normal limits.
* Symptomatic peripheral vascular disease.
* History of high dose chemotherapy with bone marrow transplant or peripheral blood stem cell transplant within the previous 2 years.
* Evidence of bleeding diathesis or coagulopathy.
* Prior treatment with an epothilone or any antiangiogenic agent.
* Concurrent nonhealing wound, ulcer, or fracture.
* Any current or history of brain and/or leptomeningeal metastases. Psychiatric disorders or other conditions rendering the participant incapable of complying with the requirements of the protocol.
* Any concurrent active malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix.
* Known allergy to any of the study drugs or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- United States (6):
  - East Valley Hematology And Oncology Medical Group, Burbank, California
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Ucsf-Comprehensive Cancer Center, San Francisco, California
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Weill Medical College Of Cornell University, New York, New York
- France (7):
  - Local Institution, Besançon
  - Local Institution, Clermont-Ferrand
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Saint-Herblain
  - Local Institution, Strasbourg
  - Local Institution, Tours
- Italy (6):
  - Local Institution, Cuneo
  - Local Institution, Meldola Fc
  - Local Institution, Milan
  - Local Institution, Modena
  - Local Institution, Napoli
  - Local Institution, Roma
- Spain (2):
  - Local Institution, Jaén
  - Local Institution, L'Hospitalet de Llobregat
- United Kingdom (4):
  - Local Institution, Chelmsford, Essex
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Merseyside, Merseyside
  - Local Institution, Nottingham, Nottinghamshire

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 136 participants enrolled in this study, 123 were randomized. Of the 13 not randomized, 11 no longer met study criteria, 1 withdrew, and 1 was found to have extensive disease. Of the 123 randomized, 122 were treated, and 1 no longer met study criteria and was never treated.
Groups:
- Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg: Ixabepilone,16 mg/m^2, administered as a 1-hour intravenous (IV) infusion on Days 1, 8, and 15 of a 28-day cycle until disease progression or unacceptable toxicity. Bevacizumab, 10 mg/kg, administered after ixabepilone as IV infusion every 2 weeks. Bevacizumab to be infused over 90 minutes for the first dose, and if well tolerated for 60 minutes, for the second dose. Then if still tolerated, over 30 minutes for subsequent infusions. Bevacizumab was to be dosed until disease progression or unacceptable toxicity.
- Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg: Ixabepilone, 40 mg/m^2, administered as a 3-hour IV infusion on Day 1 of a 21-day cycle until disease progression or unacceptable toxicity After Cycle 4, dose reduction to 32 mg/m^2 implemented for all subsequent cycles. Bevacizumab, 15 mg/kg, administered after ixabepilone as IV infusion every 3 weeks. Bevacizumab to be infused over 90 minutes for the first dose, and if well tolerated for 60 minutes, for the second dose. Then if still tolerated, over 30 minutes for subsequent infusions. Bevacizumab was to be dosed until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Started | 46 (Randomized) | 45 (Randomized) | 32 (Randomized)
Completed | 0 | 0 | 0
Not Completed | 46 | 45 | 32
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Disease progression | 23 | 23 | 15
Not completed — Maximum clinical benefit | 3 | 5 | 5
Not completed — Poor or noncompliance | 0 | 0 | 1
Not completed — Study drug toxicity | 11 | 8 | 6
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Still on treatment | 1 | 3 | 2
Not completed — Never treated | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Investigator decision | 2 | 1 | 0
Not completed — High risk of allergic reaction | 0 | 1 | 0
Not completed — Planned radiation for palliation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg | Total
Number analyzed (Participants) | 46 | 45 | 32 | 123
Age, Continuous [Median (Full Range); unit: years] | 60.0 [27.0 to 80.0] | 59.0 [37.0 to 83.0] | 59.0 [37.0 to 75.0] | 59.0 [27.0 to 83.0]
Age, Customized [Number; unit: participants]
  Younger than 65 years | 33 | 29 | 22 | 84
  >=65 years | 13 | 16 | 10 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 32 | 123
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 0 | 4
  White | 43 | 40 | 31 | 114
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Tumor Response of Partial Response (PR) or Complete Response (CR) While On-study
Description: CR=Disappearance of all clinical and radiologic evidence of target lesions; PR=At least 30% reduction in the sum of the longest diameter of all target lesions.
Time Frame: Baseline visit and then every 8 weeks to 12 months, then every 3 months until disease progression
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 46 | 45 | 32
Percentage of participants | 47.8 [32.9 to 63.1] | 71.1 [55.7 to 83.6] | 62.5 [43.7 to 78.9]

2. Secondary Outcome: Percentage of Participants With Progression-free Survival at Week 24
Description: Week 24 Progression-free Survival was defined as the number of participants who neither progressed nor died before Week 24. Computed using Kaplan-Meier estimates, only at the time of Interim Analysis, when all participants had been followed for 6 months.
Time Frame: Date of randomization to Week 24
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 46 | 45 | 32
Percentage of participants | 75 [62.37 to 87.87] | 86 [75.72 to 96.42] | 94 [85.36 to 100.00]

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to progression or to death from any cause without prior documentation of progression. Participants who did not progress or die were to be censored on the date of their last tumor assessment.
Time Frame: Date of randomization to date of progression, death, or last tumor assessment (maximum participant PFS of 29 months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 46 | 45 | 32
Months | 9.6 [6.1 to 11.7] | 11.9 [8.7 to 14.7] | 13.5 [10.0 to 18.2]

4. Secondary Outcome: Median Time to Response
Description: Time to response was defined as the time from the first dose of study therapy until measurement criteria were first met for a PR or CR, whichever was recorded first. Time to response was computed only for participants whose best response was PR or CR.
Time Frame: Date of first PR or CR assessment to date of progression, death, or last tumor assessment (maximum participant time to response of 67 weeks)
Population: Participants whose best response was CR or PR, as assessed by the investigator.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 22 | 32 | 20
Weeks | 8.2 [6.1 to 67.0] | 8.3 [5.3 to 37.9] | 8.1 [7.0 to 32.0]

5. Secondary Outcome: Median Duration of Response
Description: Duration of response was computed for participants whose best response was either PR or CR. Duration of overall response was defined as the period from the time that measurement criteria were first met for PR or CR, whichever was recorded first, until the first date of documented PD or death. Participants who neither relapsed nor died were to be censored on the date of their last tumor assessment.
Time Frame: Date of first PR or CR assessment to date of progression, death, or last tumor assessment (maximum participant duration of response of 25 weeks)
Population: Participants whose best response was CR or PR, as assessed by the investigator.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 22 | 32 | 20
Months | 10.1 [7.3 to 14.5] | 10.3 [9.0 to 14.3] | 13.1 [9.2 to 21.7]

6. Secondary Outcome: Percentage of Participants Surviving at 1 Year
Description: One year survival rates were computed using Kaplan-Meier estimates.
Time Frame: Date first participant enrolled to 1 year
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 46 | 45 | 32
Percentage of participants | 91 [82.69 to 99.42] | 89 [79.71 to 98.07] | 91 [80.53 to 100.00]

7. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs) Treatment-related SAEs, Treatment-related Adverse Events (AEs) Leading to Discontinuation, AEs Leading to Discontinuation, Treatment-related AEs
Description: An AE is any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, drug dependency or abuse; is life-threatening, an important medical event, a congenital anomaly/birth defect; requires inpatient hospitalization; or prolongs existing hospitalization. Treatment related=possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: At initiation of treatment throughout study, to a minimum of 30 days after last dose of study drug
Population: All randomized participants who received any study drug.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 45 | 45 | 32
Participants
  Deaths | 12 | 15 | 5
  SAEs | 15 | 16 | 9
  Treatment-related SAEs | 7 | 9 | 5
  Treatment-related AEs Leading to Discontinuation | 24 | 23 | 20
  AEs Leading to Discontinuation | 26 | 25 | 21
  Treatment-related AEs | 43 | 45 | 32

8. Primary Outcome: Number of Participants With Best Response As Assessed With Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Best tumor response was assessed with RECIST. Complete response (CR)=Disappearance of all evidence of target lesions; Partial response (PR)=At least 30% reduction from baseline in the sum of the longest diameter (LD) of all target lesions; Progressive disease (PD)=At least a 20% increase from baseline in the sum of LD of target lesions or the appearance of 1 or more new lesions; Stable disease (SD)=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. A response was confirmed if noted on 2 examinations at least 4 weeks apart.
Time Frame: Baseline visit and then every 8 weeks to 12 months, then every 3 months until disease progression
Population: All randomized participants
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 46 | 45 | 32
Participants
  Complete Response | 2 | 2 | 4
  Partial Response | 20 | 30 | 16
  Stable Disease | 18 | 9 | 11
  Progressive Disease | 5 | 3 | 0
  Unable to Determine | 1 | 1 | 1

9. Secondary Outcome: Number of Participants With Abnormalities in Hematology Laboratory Results by Worst Common Terminology Criteria (CTC) Grade
Description: CTC, Version 3 used to assess parameters. CTC Gr=Grade; WBC=white blood cells; ANC=absolute neutrophil count. LLN=lower level of normal. WBC Gr 1:<LLN to 3.0*10^9/L, Gr 2:<3.0 to 2.0*10^9/L, Gr 3:<2.0 to 1.0*10^9/L, Gr 4:<1.0*10^9/L; ANC Gr 1:<LLN to 1.5*10^9/L, Gr 2:<1.5 to 1.0*10^9/L, Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L; Platelet count Gr 1:LLN to 75.0*10^9/L, Gr 2:<75.0 to 50.0*10^9/L, Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L; Hemoglobin Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL.
Time Frame: At initiation of treatment and throughout study, to a minimum of 30 days after last dose of study drug. Laboratory tests performed within 72 hours before start of each cycle
Population: All randomized participants who received any study drug.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 45 | 45 | 32
Participants
  White blood cells (WBC) (Grade 1) | 11 | 12 | 12
  WBC (Grade 2) | 14 | 12 | 11
  WBC (Grade 3) | 1 | 14 | 3
  WBC (Grade 4) | 2 | 4 | 0
  Absolute neutrophil count (ANC) (Grade 1) | 10 | 4 | 6
  ANC (Grade 2) | 9 | 10 | 13
  ANC (Grade 3) | 5 | 17 | 6
  ANC (Grade 4) | 2 | 10 | 1
  Platelet count (Grade 1) | 4 | 15 | 3
  Platelet count (Grade 2) | 1 | 1 | 0
  Platelet count (Grade 3) | 0 | 0 | 0
  Platelet count (Grade 4) | 2 | 1 | 0
  Hemoglobin (Grade 1) | 21 | 20 | 17
  Hemoglobin (Grade 2) | 3 | 4 | 3
  Hemoglobin (Grade 3) | 1 | 3 | 2
  Hemoglobin (Grade 4) | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With Abnormalities in Liver Function by Worst CTC Grade
Description: ULN=Upper limit of normal.ALT Gr 1:>ULN to 2.5*ULN, Gr 2: >2.5 to 5.0*ULN, Gr 3: >5.0 to 20.0*ULN, Gr 4: >20.0*ULN; AST Gr 1: >ULN to 2.5*ULN, Gr 2: >2.5 to 5.0*ULN, Gr 3: >5.0 to 20.0*ULN, Gr 4: >20.0*ULN; ALP Gr 1:>ULN to 2.5*ULN, Gr 2: >2.5 to 5.0*ULN, Gr 3: >5.0 to 20.0*ULN, Gr 4: >20.0*ULN; Total bilirubin Gr 1: >ULN to 1.5*ULN, Gr 2: >1.5 to 3.0*ULN, Gr 3: >3.0 to 10.0*ULN, Gr 4: >10.0*ULN.
Time Frame: as for outcome 9
Population: All randomized participants who received any study drug and had samples available.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 43 | 44 | 32
Participants
  Alanine aminotransferase (ALT) (Grade 1) | 18 | 13 | 13
  ALT (Grade 2) | 2 | 4 | 3
  ALT (Grade 3) | 1 | 0 | 0
  ALT (Grade 4) | 0 | 0 | 0
  AST (Grade 1) | 20 | 18 | 15
  AST (Grade 2) | 1 | 1 | 1
  AST (Grade 3) | 1 | 0 | 0
  AST (Grade 4) | 0 | 0 | 0
  Alkaline phosphatase (ALP) (Grade 1) | 8 | 11 | 12
  ALP (Grade 2) | 0 | 3 | 0
  ALP (Grade 3) | 0 | 0 | 1
  ALP (Grade 4) | 0 | 0 | 0
  Total bilirubin (Grade 1) | 3 | 3 | 2
  Total bilirubin (Grade 2) | 2 | 0 | 1
  Total bilirubin (Grade 3) | 0 | 0 | 0
  Total bilirubin (Grade 4) | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Abnormalities in Renal Function by Worst CTC Grade
Description: Creatine Gr 1: >ULN to 1.5*ULN, Gr 2: 1.5 to 3.0*ULN, Gr 3: >3.0 to 6.0*ULN, Gr 4: >6.0*ULN.
Time Frame: as for outcome 9
Population: All randomized participants who received any study drug and had samples available.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Number analyzed (Participants) | 44 | 44 | 32
Participants
  Creatinine (Grade 1) | 5 | 3 | 3
  Creatinine (Grade 2) | 3 | 1 | 0
  Creatinine (Grade 3) | 0 | 0 | 0
  Creatinine (Grade 4) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Continuously from first to last dose of study drug (24 weeks)and within 30 days following last dose.
Groups:
- Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg: Ixabepilone,16 mg/m^2, administered as a 1-hour intravenous (IV) infusion on Days 1, 8, and 15 of a 28-day cycle until disease progression or unacceptable toxicity. Bevacizumab, 10 mg/kg, administered after ixabepilone, as IV infusion every 2 weeks. Bevacizumab to be infused over 90 minutes for the first dose, and if well tolerated for 60 minutes, for the second dose. Then if still tolerated, over 30 minutes for subsequent infusions. Bevacizumab was to be dosed until disease progression or unacceptable toxicity.
- Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg: Ixabepilone, 40 mg/m^2, administered as a 3-hour IV infusion on Day 1 of a 21-day cycle until disease progression or unacceptable toxicity. After Cycle 4, dose reduction to 32 mg/m^2 implemented for all subsequent cycles. Bevacizumab, 15 mg/kg, administered after ixabepilone, as IV infusion every 3 weeks. Bevacizumab to be infused over 90 minutes for the first dose, and if well tolerated for 60 minutes, for the second dose. Then if still tolerated, over 30 minutes for subsequent infusions. Bevacizumab was to be dosed until disease progression or unacceptable toxicity.
Arm/Group | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 15/45 | 16/45 | 9/32
Other Adverse Events (participants affected / at risk) | 45/45 | 45/45 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg (N=45) | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg (N=45) | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg (N=32)
Blood creatinine increased (Investigations) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 2 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Complicated migraine (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Bacteroides infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hernia (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 16 mg/m^2 + Bevacizumab, 10 mg/kg (N=45) | Ixabepilone, 40 mg/m^2 + Bevacizumab, 15 mg/kg (N=45) | Paclitaxel, 90 mg/m^2 + Bevacizumab, 10 mg/kg (N=32)
Dry eye (Eye disorders) | 0 | 1 | 2
Vision blurred (Eye disorders) | 3 | 0 | 3
Weight decreased (Investigations) | 7 | 9 | 3
Weight increased (Investigations) | 3 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 3
Tachycardia (Cardiac disorders) | 0 | 1 | 3
Flushing (Vascular disorders) | 1 | 0 | 2
Hot flush (Vascular disorders) | 3 | 2 | 5
Haemorrhage (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 4 | 1 | 1
Hypertension (Vascular disorders) | 14 | 22 | 10
Anxiety (Psychiatric disorders) | 5 | 8 | 4
Insomnia (Psychiatric disorders) | 5 | 9 | 6
Depression (Psychiatric disorders) | 3 | 3 | 3
Depressed mood (Psychiatric disorders) | 1 | 1 | 2
Hypersensitivity (Immune system disorders) | 3 | 2 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 17 | 15 | 14
Lethargy (Nervous system disorders) | 3 | 2 | 3
Migraine (Nervous system disorders) | 1 | 0 | 2
Sciatica (Nervous system disorders) | 2 | 1 | 2
Dizziness (Nervous system disorders) | 4 | 2 | 4
Dysgeusia (Nervous system disorders) | 9 | 9 | 4
Somnolence (Nervous system disorders) | 0 | 1 | 2
Dysaesthesia (Nervous system disorders) | 3 | 2 | 2
Paraesthesia (Nervous system disorders) | 11 | 11 | 8
Hypoaesthesia (Nervous system disorders) | 2 | 3 | 2
Neuropathy peripheral (Nervous system disorders) | 12 | 14 | 14
Peripheral motor neuropathy (Nervous system disorders) | 4 | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 19 | 12
Nausea (Gastrointestinal disorders) | 18 | 14 | 12
Vomiting (Gastrointestinal disorders) | 16 | 6 | 13
Diarrhea (Gastrointestinal disorders) | 27 | 14 | 18
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 2
Gastritis (Gastrointestinal disorders) | 3 | 1 | 1
Toothache (Gastrointestinal disorders) | 3 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 3
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 4 | 10 | 5
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 20 | 12 | 10
Hemorrhoids (Gastrointestinal disorders) | 4 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 11 | 11 | 7
Gingival bleeding (Gastrointestinal disorders) | 4 | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7 | 1
Vertigo (Ear and labyrinth disorders) | 6 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 4 | 2 | 7
Sinusitis (Infections and infestations) | 2 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2
Laryngitis (Infections and infestations) | 0 | 3 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 2
Pharyngitis (Infections and infestations) | 1 | 2 | 3
Folliculitis (Infections and infestations) | 1 | 4 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 2
Skin infection (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 4 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 3 | 5
Vaginal infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2
Dysuria (Renal and urinary disorders) | 5 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 10 | 9 | 4
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 7 | 10 | 8
Rash (Skin and subcutaneous tissue disorders) | 8 | 4 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 22 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 4 | 6
Erythema (Skin and subcutaneous tissue disorders) | 2 | 6 | 7
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 10 | 8 | 15
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 12 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 9 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 6 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 10 | 9
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 8 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 | 17 | 21
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Pain (General disorders) | 2 | 3 | 2
Fatigue (General disorders) | 13 | 9 | 10
Pyrexia (General disorders) | 7 | 10 | 9
Asthenia (General disorders) | 20 | 23 | 13
Chest pain (General disorders) | 4 | 3 | 2
Chest discomfort (General disorders) | 1 | 0 | 2
Edema peripheral (General disorders) | 5 | 8 | 4
Mucosal inflammation (General disorders) | 7 | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period of 60 days or less from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.